CLINICAL TRIAL: NCT03154658
Title: Serratus Anterior Plane Block: Sub-Serratus vs Supra-Serratus Plane Block for Pain Control in Patients Undergoing Mastectomy
Brief Title: Serratus Anterior Plane Block in Patients Undergoing Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Machi, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 122016-011
Record Dates: First submitted 2017-05-03; First posted 2017-05-16 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Pain, Post-operative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized interventional prospective model to investigate effect of block placement in two treatment arms. Opioid consumption in the first 24 hours after the operation will be main outcome variable.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub-serratus regional block (Experimental): A regional block using of ropivacaine 0.35% (30 mL will be used per side in patients weighing over 60 kg and 20 mL will be used in patients weighing less than 60 kg) will be administered to the injection site deep to the serratus anterior muscle.
  Interventions: Drug: Ropivacaine 0.35%
- Supra-serratus regional block (Active Comparator): A regional block using of ropivacaine 0.35% (30 mL will be used per side in patients weighing over 60 kg and 20 mL will be used in patients weighing less than 60 kg) will be administered to the injection site superficial to the serratus anterior muscle.
  Interventions: Drug: Ropivacaine 0.35%

INTERVENTIONS:
Drug: Ropivacaine 0.35% — The serratus plane block is used to supplement the pain management of a patient receiving a surgical procedure of the chest wall or breast.
  Other Names: Ropivacaine

SUMMARY:
This is a randomized, interventional prospective study. Patients (n=66) undergoing mastectomies with or without tissue expander will be randomized to receive a supra-serratus or sub-serratus regional plane block prior to surgery. The main effect to be measured is total opioid consumption 24 hours after the operation. Secondary endpoints include measuring a change between pre-and post-operative pain scores, patient satisfaction of pain control during first 24 hours after the operation, presence of postoperative nausea and vomiting, duration of sleep on first postoperative night, and block performance time and length of stay, between the two treatment arms.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two groups: the supra-serratus anterior plane block (depositing local anesthetic superficial to the serratus anterior muscle) or the sub-serratus anterior plane block (depositing local anesthetic deep to the serratus anterior muscle). Randomization will be performed using a computer generated randomization program. The results of the randomization will be revealed to the physician performing the block just prior to its performance. The site of the block will be marked and a safety timeout will be performed with the block nurse, regional anesthesiologist, and patient present and participating.

Once the above is completed, patients will receive a pre-operative ultrasound-guided single-injection serratus anterior plane block using either the supra-serratus or sub-serratus techniques according to their randomization. The block nurse will record the time when the timeout is performed, the "needle insertion" time when the block needle enters the skin, and the "block complete" time when the needle exits the skin. If the block is bilateral, the block nurse will record the time when the timeout is performed, then will record two sets of "needle in" times and "needle out" times, one for each side. In the case of a bilateral block, the same method of serratus anterior plane block will be utilized for both sides.

After the block, the patient will proceed to surgery. The operating room anesthesia team will be notified that the patient received a serratus anterior plane block. An appropriate multimodal general anesthetic will be employed at the operating room anesthesiologist's discretion. Upon completion of the surgery and emergence from general anesthesia, the patient will be seen by study personnel in the Post Anesthesia Care Unit and pain will be evaluated using a 0-10 Likert scale (0=no pain, 10= worst imaginable pain) about 1 hour post-operatively. Pain will be evaluated again by study personnel using the same scale on post-operative day #1, about 24 hours after initial block placement. If the patient is discharged home prior to the post-operative day #1 assessment, a phone interview will be performed 24 hours following the block to evaluate the post-operative day #1 scores and monitor for adverse events. Additional pain scores will be documented in the electronic medical record by nursing staff per protocol, and will be collected by study personnel.

During the intraoperative and post-operative period, the patient will continue to receive an appropriate multimodal analgesic regimen as necessary to adequately control the pain. No pain control method will be withheld from the patient as a result of participating in the study.

Patient satisfaction scores will also be used as a measure to evaluate quality of perioperative pain management. These scores will be assessed on post-operative day #1 on a scale of 1 to 5 (Poor=1, Fair=2, Good=3 Very good=4, Excellent=5).

During follow-up on post-operative day #1, the patients will also be asked for an estimate on duration and quality of sleep to help assess their general comfort level during their first post-operative night.

During the routine post-operative visit, an assessment of post-operative nausea and vomiting will be made by asking the patient directly. Chart review looking for post-operative antiemetic usage will also be evaluated to assess the presence of post-operative nausea and vomiting.

The decision as to whether or not to perform a serratus anterior plane block (SAPB) will be made independent from the introduction of the patient to the study. Therefore, the patient's choice to receive a SAPB will not be affected by the introduction of the study or their desire to participate in a clinical investigation. A multimodal intraoperative anesthetic technique will be employed for all patients, and post-operative pain control will be managed by the patient's primary surgical team.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years or older
2. Individuals undergoing either a mastectomy or mastectomy with tissue expander for which the anesthetic plan includes a serratus anterior plane block.

Exclusion Criteria:

1. Any known sensory deficit of the anterolateral chest wall.
2. Any local disorder of the skin or otherwise where blockade is to be performed which would prevent safe performance of the block
3. Pregnancy
4. American Society of Anesthesiology classification greater than 3
5. Allergy to amide local anesthetic medications
6. Chronic pain conditions
7. Preoperative opioid use greater than 20 oral morphine equivalents per day
8. Any coagulation abnormality which would be a contraindication for block placement
9. Preoperative chronic renal dysfunction requiring renal replacement therapy or a serum creatinine greater than 1.4 mg/dL
10. Body mass index >50
11. Incarceration
12. Inability to understand study procedures including inability to understand the English language
13. Inability to provide adequate informed consent
14. Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Machi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Centers, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards JT, Langridge XT, Cheng GS, McBroom MM, Minhajuddin A, Machi AT. Superficial vs. deep serratus anterior plane block for analgesia in patients undergoing mastectomy: A randomized prospective trial. J Clin Anesth. 2021 Dec;75:110470. doi: 10.1016/j.jclinane.2021.110470. Epub 2021 Aug 5. PMID 34364099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Women over the age of 18 who underwent a mastectomy, either unilateral or bilateral, with or without tissue expander placement, and with or without axillary node dissection were recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (14.2) | 52.0 (11.0) | 53.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (6.4) | 30.2 (10.5) | 29.0 (8.7)
Intraoperative length [Mean (Standard Deviation); unit: minutes] | 321.6 (110.1) | 323.0 (114.7) | 322.3 (111.6)
Tissue expander placement [Number; unit: participants] | 24 | 27 | 51
Axillary node dissection [Number; unit: participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Measures number of milligrams morphine equivalents each subject receives
Time Frame: 24 hours post block
Measure: Median (Inter-Quartile Range); unit: milligrams oral morphine equivalent
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
milligrams oral morphine equivalent | 113.5 [86.5 to 176.2] | 147 [126.5 to 227.0]

2. Secondary Outcome: Maximum Post-operative Pain Score
Description: Measures the change in pain scores on a 0-10 Numeric Rating Scale where 0 is no pain and 10 is the maximum pain.
Time Frame: 24 hours post block
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
units on a scale | 5.2 (4.4) | 5.9 (5.2)

3. Secondary Outcome: Patient Satisfaction Scale
Description: Pain satisfaction with regards to post-operative pain management within the first 24 hours post op on a 1-5 Likert scale of (1 poor, 2 fair, 3 good, 4 very good, 5 excellent).
Time Frame: 24 hours post block
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
units on a scale | 3.62 (1.01) | 3.24 (0.91)

4. Secondary Outcome: Number of Participants With Nausea/Vomiting
Description: Measures the type and frequency of anti-emetics subjects receive
Time Frame: 24 hours post block
Measure: Number; unit: participants
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
participants | 14 | 15

5. Secondary Outcome: Length of Stay
Description: Measures total number of days subject is hospitalized, including day of surgery
Time Frame: 10 Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
days | 2 [1 to 2] | 2 [1 to 2]

6. Secondary Outcome: Sleep Duration Night of Postoperative Day 0
Description: Measures the total duration of sleep in minutes that subjects report sleeping on the night after surgery between postoperative days 0 and 1
Time Frame: 24 hours post block
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
minutes | 315 (114) | 276 (80.4)

7. Secondary Outcome: Block Performance Time
Description: Measures total time for block to take effect
Time Frame: Time from procedure needle insertion until needle removal, estimate less than 5 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
Number analyzed (Participants) | 32 | 32
minutes | 8 [6 to 10] | 7.5 [5.5 to 11.5]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Sub-serratus Regional Block | Supra-serratus Regional Block
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 14/32 | 15/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-serratus Regional Block (N=32) | Supra-serratus Regional Block (N=32)
Nausea in first 24 hours after surgery (Gastrointestinal disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT03154658/Prot_SAP_000.pdf